CLINICAL TRIAL: NCT03585296
Title: A Phase 2 Safety Study of ATI-502 Topical Solution in Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: A Study of ATI-502 Topical Solution for the Treatment of Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATI-502-AD-201
Record Dates: First submitted 2018-06-25; First posted 2018-07-13 (Actual); Results first posted 2020-02-06 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2018-08

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ATI-502 (Experimental): ATI-502 topical solution applied daily for four weeks.
  Interventions: Drug: ATI-502

INTERVENTIONS:
Drug: ATI-502 — Topical Solution

SUMMARY:
This is an open label, multicenter study designed to evaluate the safety and tolerability of ATI-502 Topical Solution in male and female subjects with moderate or severe atopic dermatitis (AD). Subjects will be required to apply ATI-502 study medication to their identified AD treatment areas. All subjects will be required to complete a safety follow up visit 4 weeks post last study medication application

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-nursing female subjects ≥ 18 years old at the time of informed consent.
2. Subject must have diagnosis of AD.
3. Subject must have a diagnosis of moderate or severe AD for a period of ≥6 months prior to the first dose of study medication.
4. Body surface area involvement must be between 2-20%.
5. Subject must have an absolute neutrophil count and a platelet count within normal range.
6. Subject must be willing to refrain from excess of sun exposure.
7. Subjects must refrain from participating in strenuous exercise that would cause profuse sweating for a period of 6 hours after each treatment application with ATI-502.
8. Be in good general health and free of any known disease state or physical condition which, in the investigator's opinion, might impair evaluation of the subject or which might expose the subject to an unacceptable risk by study participation.
9. If a woman of childbearing potential (WOCBP), must have a negative serum pregnancy test at Screening and a negative urine pregnancy test at Baseline and agree to: use a highly effective method of birth control for the duration of the study; not be planning a pregnancy during the study duration and use contraception for 30 days after last application of study medication.
10. Sexually active male subjects must agree to use a barrier method of contraception from the first application of study medication to at least 30 days after the last application of study medication.

Exclusion Criteria:

1. Subject has any signs or symptoms associated with AD therapy which, in the investigator's opinion, might impair evaluation of the AD or which exposes the subject to unacceptable risk by study participation.
2. Subjects unable to complete the required washout periods. Use of prescription moisturizers within 7 days of Visit 1.
3. Subject has used any emollients/moisturizers on the planned treatment area (s) within 4 hours of Visit 1.
4. Subject has clinically infected AD.
5. Subject is currently using an oral H1 antihistamines (e.g. diphenhydramine, terfenadine) UNLESS the subject is on a stable dose for at least 14 days prior to Visit 1.
6. Clinically significant laboratory abnormalities at Visit 1 that, in the opinion of the Investigator, would make the subject a poor candidate for the study.
7. History of, or current, severe, progressive or uncontrolled renal, hepatic, gastrointestinal, pulmonary, cardiovascular, genitourinary (renal disease) or hematological disease, neurologic or cerebral disorders, infectious disease or coagulation disorders that, as determined by the Investigator, would preclude participation in and completion of study assessments.
8. History of, current or suspected systemic or cutaneous malignancy and /or lymphoproliferative disease, other than subjects with: a history of adequately treated and well healed and completely cleared non-melanoma skin cancers (basal or squamous cell carcinoma) treated successfully at least 1 year prior to study entry with no evidence of disease.
9. Evidence of active or latent bacterial (including tuberculosis) or viral infections at the time of enrollment or history of incompletely treated or untreated tuberculosis. Subjects who have completed therapy for latent tuberculosis may participate.
10. History of a serious local infection (e.g., cellulitis, abscess) or systemic infection including but not limited to a history of treated infection (e.g., pneumonia, septicemia) within 3 months prior to Visit 2. Subjects on an antibiotic for a non-serious, acute local infection must complete the course prior to enrollment into the study.
11. Positive serological test for HIV(antibody), HCV (antibody), or HepB (HBsAg). Subjects with herpes zoster or cytomegalovirus (CMV) that resolved less than 2 months before study enrollment. Subjects with a history of frequent outbreaks of Herpes Simplex Virus (defined as 4 or more outbreaks a year).
12. Screening ECG findings of:

    1. QTcF >450msec for males or >470msec for females.
    2. Heart rate < 45 or > 100 beats/minutes (inclusive).
    3. Rhythm disturbance other than sinus arrhythmia or ectopic supraventricular rhythm (ectopic atrial rhythm).
    4. Conduction disturbance including PR >240msec, pre-excitation (delta wave and PR <120msec), second degree or higher AV block.
    5. Acute or chronic signs of ischemia.
    6. Left Bundle Branch Block.
    7. Prior myocardial infarction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judy Schynder, MBA, Study Chair — Aclaris Therapeutics
Locations (6):
- United States (6):
  - Aclaris Investigational Site, Encinitas, California
  - Aclaris Investigator Site, San Diego, California
  - Aclaris Investigator Site, Fridley, Minnesota
  - Aclaris Investigational Site, Bexley, Ohio
  - Aclaris Investigational Site, Portland, Oregon
  - Aclaris Investigator Site, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ATI-502: 0.46% Solution applied twice a day for 28 days
Period: Overall Study
Arm/Group | ATI-502
Started | 22
Completed | 17
Not Completed | 5
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | ATI-502
Number analyzed (Participants) | 22
Age, Customized [Count of Participants; unit: Participants]
  < 35 years of age | 11
  >/= 35 years of age | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 2
  White | 13
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects withTreatment-Emergent Adverse Events (Safety and Tolerability)
Description: Treatment emergent adverse events (TEAEs)graded on a 3 point scale of mild, moderate or severe
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-502
Number analyzed (Participants) | 22
Participants | 7

ADVERSE EVENTS:
Time Frame: 56 days
Description: An AE is the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered casually related to the product. In clinical studies, an AE can include an undesirable medical condition occurring at any time, including baseline or washout periods, even if no study treatment has been administered.
Arm/Group | ATI-502
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 1/22
Other Adverse Events (participants affected / at risk) | 7/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ATI-502 (N=22)
Cellulitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ATI-502 (N=22)
Chalazion (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Gastroenteritis viral (Gastrointestinal disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-17): https://cdn.clinicaltrials.gov/large-docs/96/NCT03585296/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-14): https://cdn.clinicaltrials.gov/large-docs/96/NCT03585296/SAP_001.pdf